CLINICAL TRIAL: NCT04490096
Title: Multimodal Imaging Outcome Measures for ALS (Image ALS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding issues.
Sponsor: University of Pennsylvania (Other)
Collaborators: Biogen (Industry); University of Miami (Other); University of Kansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 834366
Record Dates: First submitted 2020-06-24; First posted 2020-07-28 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: ALS
MeSH Terms: interventions — (methyl-(11)C)N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [11C]-PBR28 ALS (Other): Neuroinflammatory pathways have been implicated in a variety of neurodegenerative disorders including amyotrophic lateral sclerosis (ALS), but the vast majority of this evidence is from animal or ex vivo human studies. In vivo measurement of the 18 kDa translocator protein (TSPO) has become possible with [11C]-PBR28 PET imaging. Briefly, TSPO expression is increased when microglial are activated. Cross-sectional studies have demonstrated that [11C]-PBR28 uptake is elevated in ALS compared to controls, is correlated with upper motor neuron severity, and that microglial activation is associated with more severe upper motor neuron disease and faster disease progression. We are only aware of a single 6-month study of 10 patients evaluating longitudinal change of [11C]-PBR28 in ALS. We hypothesize that we will observe increased [11C]-PBR28 uptake over a 6-month period in motor cortex and prefrontal cortex in ALS. This portion of the study will be performed at UPenn only.
  Interventions: Drug: [11C]-PBR28

INTERVENTIONS:
Drug: [11C]-PBR28 — A dose of ≤ 20 mCi (approximate range for most studies is anticipated to be 5-20 mCi) of [11C]-PBR28 will be administered by IV injection to the patient under the direct supervision of a Nuclear Medicine Authorized User. A lesser activity may be injected if, in the opinion of a nuclear medicine authorized user complete imaging data could be generated.
  Subjects will undergo an approximately 90 minute dynamic PET/CT scan over the brain starting at approximately the same time as the [11C]-PBR-28 injection. Scans will be acquired using a Philips PET/CT time-of-flight Ingenuity scanner (Philips Healthcare, Cleveland, OH, USA). At the end of the dynamic imaging the participant will be allowed to get off the scanner.

SUMMARY:
The primary aim of this study is to determine whether longitudinal neuroimaging acquired across multiple research and clinical centers is a feasible biomarker to use as an outcome measure for clinical trials in amyotrophic lateral sclerosis (ALS)

DETAILED DESCRIPTION:
ALS is a progressive neurodegenerative disorder that manifests with extensive clinical heterogeneity, including variable degrees of upper motor neuron (UMN) and lower motor neuron (LMN) impairment. While ALS is classically defined as a neuromuscular disorder, approximately 15% of individuals also develop cognitive and/or behavioral dysfunction of the frontotemporal variety, ranging in severity from ALS with cognitive or behavior impairment to a frank form of dementia consistent with FTD2

* Recent consensus criteria capture this heterogeneity by defining these conditions together as amyotrophic lateral sclerosis frontotemporal spectrum disorder (ALS-FTSD)3
* There are emerging and in-progress interventional clinical trials underway that aim to arrest ALS and/or FTD disease progression; however, there are limited objective and quantitative biomarkers to directly track disease progression during life. Multi-modal neuroimaging provides an ideal candidate biomarker for clinical trials because ALS-FTSD affects a distributed neuroanatomic network and we can reliably measure neurodegeneration of grey matter (GM) and arterial spin labeling based perfusion MRI (pMRI) measurements of cerebral blood flow (CBF). However, there are many unaddressed technical challenges associated with measuring disease progression using neuroimaging techniques in a multi-center setting. The overall aim of this protocol is to leverage a team science approach to develop disease-specific candidate neuroimaging outcome measures for ALS-FTSD clinical trials.

ELIGIBILITY:
Inclusion criteria for participants in PET sub-study (Penn Only):

1. Enrolled in the MRI study at Penn.
2. Willing to participate in a 30 minute [18F]-FDG and 1.5 hour [11C]-PBR28 PET scan within 15 days baseline and longitudinally at the 3-month and 6-month follow-up visits, if able.

Exclusion criteria for PET sub-study participants:

1. Females who are pregnant at the time of study visits will not be eligible for the PET sub-study; urine or serum pregnancy test will be performed in women of child-bearing potential at each of the baseline, 3-month, and 6-month study visit.
2. Homozygous genotype for the threonine-associated substitution allele (A) in the rs6971 polymorphism.
3. Blood glucose less than or equal to 250 mg/dl, or at the discretion of the authorized user

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Volume measurement (cubic mm) of brain regions using MRI | Change from baseline volume measurement (cubic mm) at 6 months
  Volume measurement (cubic mm) of brain regions using MRI for ALS patients and healthy controls.
Volume measurement (cubic mm) of brain regions using MRI | Change from baseline volume measurement (cubic mm) at 12 months
  Volume measurement (cubic mm) of brain regions using MRI for ALS patients and healthy controls.
Thickness measurement (mm) of brain regions using MRI | Change from baseline thickness measurement (mm) at 6 months
  Thickness measurement (mm) of brain regions using MRI in ALS patients and healthy controls.
Thickness measurement (mm) of brain regions using MRI | Change from baseline thickness measurement (mm) at 12 months
  Thickness measurement (mm) of brain regions using MRI in ALS patients and healthy controls.
Cerebral blood flow measurement (mL of blood/100g per minute) of brain regions using MRI | Change from baseline cerebral blood flow measurement (mL of blood/100g per minute) at 6 months
  Determine whether MRI is a feasible for measuring longitudinal change comparing ALS patients relative to healthy controls. ALS will have increased rate of hyperperfusion, reflected by reduced cerebral blood flow (mL of blood/100g per minute), in the motor cortex and frontal cortex brain regions relative to healthy controls.
Cerebral blood flow measurement (mL of blood/100g per minute) of brain regions using MRI | Change from baseline cerebral blood flow measurement (mL of blood/100g per minute at 12 months
  Determine whether MRI is a feasible for measuring longitudinal change comparing ALS patients relative to healthy controls. ALS will have increased rate of hyperperfusion, reflected by reduced cerebral blood flow (mL of blood/100g per minute), in the motor cortex and frontal cortex brain regions relative to healthy controls.

SECONDARY OUTCOMES:
[18F]-FDG signal measurement (standard uptake volume or SUV) in brain regions using PET scan | Change from baseline [18F]-FDG signal measurement (standard uptake volume or SUV) at 3 months
  [18F]-FDG signal measurement (Standard Uptake Value or SUV) of [18F]-FDG PET for ALS patients at PENN only.
[18F]-FDG signal measurement (standard uptake volume or SUV) in brain regions using PET scan | Change from baseline [18F]-FDG signal measurement (standard uptake volume or SUV) at 6 months
  [18F]-FDG signal measurement (Standard Uptake Value or SUV) of [18F]-FDG PET for ALS patients at PENN only.
[11C]-PBR28 signal measurement (standard uptake volume or SUV) in brain regions using PET scan | Change from baseline [11C]-PBR28 signal measurement (standard uptake volume or SUV) at 3 months
  [11C]-PBR28 signal measurement (Standard Uptake Value or SUV) of [11C]-PBR28 PET for ALS patients at PENN only.
[11C]-PBR28 signal measurement (standard uptake volume or SUV) in brain regions using PET scan | Change from baseline [11C]-PBR28 signal measurement (standard uptake volume or SUV) at 6 months
  [11C]-PBR28 signal measurement (Standard Uptake Value or SUV) of [11C]-PBR28 PET for ALS patients at PENN only.

CONTACTS AND LOCATIONS:
Overall Officials: Corey McMillan, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No